CLINICAL TRIAL: NCT05632731
Title: Comparison of Clinical Outcomes in Fresh Cycle With Single Blastocyst Stage and Double Cleavage-stage Embryos: a Single-center, Non-blind, Randomized Controlled Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Collaborators: ORGANON (SHANGHAI) PHARMACEUTICAL TECHNOLOGY CO., LTD. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-20220201-R
Record Dates: First submitted 2022-11-20; First posted 2022-12-01 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Double Cleavage-stage Embryos transfer (Other): In group A, two embryos at cleavage stage were transplanted on the third day after oocyte retrieval.
  Interventions: Procedure: double cleavage-stage or single blastocyst stage embryos transfer
- Single Blastocyst Stage Embryos transfer (Other): Group B was graded by Gardner blastocyst grading method, and one blastocyst was transplanted on the 5th or 6th day after oocyte retrieval.
  Interventions: Procedure: double cleavage-stage or single blastocyst stage embryos transfer

INTERVENTIONS:
Procedure: double cleavage-stage or single blastocyst stage embryos transfer — Infertile women requesting in vitro fertilization treatment were randomly assigned to undergo transfer of either two cleavage-stage embryos or a single blastocyst-stage embryo.

SUMMARY:
In traditional assisted reproductive technology (ART), choosing multiple embryo transfer to get a high clinical pregnancy rate while increasing the risk of multiple pregnancies. Research showed that the single-cleavage embryo transfer could not simultaneously meet the dual requirements of maintaining pregnancy rate and reducing the multiple pregnancy rate.The purpose of this study was to observe the clinical outcome between double cleavage embryo transfers and single blastocyst transfers in fresh cycle through RCT study with GnRH antagonist protocol.

DETAILED DESCRIPTION:
In traditional assisted reproductive technology (ART), choosing multiple embryo transfer to get a high clinical pregnancy rate while increasing the risk of multiple pregnancies. Research showed that in the fresh cleavage embryo transfer cycle, the clinical pregnancy rate increased with the increase of the number of high-quality embryos transferred, and so did the multiple pregnancy rate, suggesting that the single-cleavage embryo transfer could not simultaneously meet the dual requirements of maintaining pregnancy rate and reducing the multiple pregnancy rate. Compared with the embryo at cleavage stage, blastocyst culture is a process of survival of the fittest, which is physiologically more synchronized with endometrial development and can improve embryo implantation rate.

The existing clinical research analysis is mostly limited to the down-regulating regimen, while the RCT study of high-quality with GnRH antagonist protocol is few. Therefore, the purpose of this study was to observe the clinical outcome between double cleavage embryo transfers and single blastocyst transfers in fresh cycle through RCT study with GnRH antagonist protocol.

ELIGIBILITY:
Inclusion Criteria:

1. patients with a diagnosis of primary or secondary infertility with a clinical indication for IVF/intracytoplasmic sperm injection (ICSI)
2. under 38 years of age
3. number of AFC≥6, AMH>1.1ng/ml
4. no adverse factors of fresh embryo transplantation (evaluation by an experienced reproductive physician)
5. number of available embryos(day 3)≥4
6. informed consent

Exclusion Criteria:

1. PGT
2. with adenomyosis, endometrial compression by uterine fibroids, intrauterine adhesion, endometrial polyps and other factors unsuitable for fresh cycle transplantation

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1236 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
live birth rate per fresh transfer | 2 year
  live birth, which was defined as the presence of a live fetus (or feti) after the 24th week of gestational age